CLINICAL TRIAL: NCT06857786
Title: Open Label, Multicenter, Phase Ib Trial of CT041, Claudin 18.2 Specific CAR T Cell Therapy As a Consolidation Therapy After Adjuvant Therapy for Resected Gastric or Gastroesophageal Junction Adenocarcinoma Patients
Brief Title: Postoperative Adjuvant Therapy for CT041 Gastric or Gastroesophageal Junction (G/GEJ) Adenocarcinoma Patients
Acronym: CT041-CG4010
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT041-CG4010
Record Dates: First submitted 2025-01-08; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Gastric Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Drug: CT041 autologous CAR T-cell injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1b, open-label, single-arm trial (Experimental): Drug: CT041 autologous CAR T-cell injection
  Interventions: Drug: Drug: CT041 autologous CAR T-cell injection

INTERVENTIONS:
Drug: Drug: CT041 autologous CAR T-cell injection — The planned dose of satri-cel in this trial was 2.5 × 108 cells, single infusion. The trial will start with a safety run-in phase, which is defined from the day of infusion to the 28th day after infusion for the first 6 participants. The type, grade, incidence rate, and outcome of adverse events during the safety run-in phase will be summarized and assessed by the investigator and collaborator (CARsgen Therapeutics Co., Ltd). The investigator and collaborator could discuss and assess whether the lower or higher doses should be explored based on the based on the safety and tolerability, cellular metabolic characteristics, and benefit-risk profile. If no dose adjustment is required, satri-cel dose will continue to be 2.5 × 108 cells for the rest of the participants.

SUMMARY:
To evaluate the safety and tolerability of satri-cel as consolidation therapy after postoperative adjuvant therapy in patients with resected gastric or gastroesophageal junction (G/GEJ) adenocarcinoma

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate the safety and tolerability of satri-cel as consolidation therapy after postoperative adjuvant therapy in patients with G/GEJ adenocarcinoma. The primary endpoint is the frequency, type, severity and outcome of AE/SAE/AESI, which is the routine assessment indicators for evaluating the safety and tolerability of the investigational product in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must have voluntarily signed the informed consent form (ICF) and be willing to comply with all trial procedures.

  2. Must be 18 -75 years old (inclusive), male or female. 3. Pathologically confirmed diagnosis of gastric/gastroesophageal junction (G/GEJ) adenocarcinoma.

  4. Must have CLDN18.2-positive tumor expression as determined by immunohistochemistry (IHC), defined as CLDN18.2 staining intensity ≥ 1+ in at least 70% of tumor cells.

  5. Must have undergone D2 gastrectomy and achieved R0 resection. 6. Must have pathological stage (y)pT4aN+ or (y)pT4bNany) according to the American Joint Committee on Cancer (AJCC) TNM Staging Classification (8th ed., 2017).

  7. Must have received full cycles of standard adjuvant chemotherapy according to treatment guidelines. Standard adjuvant chemotherapy allowed in this trial includes FLOT(docetaxel + oxaliplatin + fluorouracil), CapeOX (oxaliplatin + capecitabine), and FOLFOX(oxaliplatin + fluorouracil).
  1. Neoadjuvant chemotherapy is allowed.
  2. Participants who are deemed intolerable or medically improper to complete the full cycles of adjuvant chemotherapy or not beneficial as determined by the investigator could be eligible after discussing with the medical monitor.

     8. Must have no evidence of recurrent or metastatic G/GEJ adenocarcinoma. 9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (within 7 days before leukapheresis).

     10. Sufficient venous access for leukapheresis collection and no other contraindications to leukapheresis.

     11. Laboratory results within 7 days before leukapheresis must meet the following criteria (Retesting once within one week is permitted. it will be considered a screening failure if retest still not meets the criteria): 12. Women of childbearing potential (WOCBP) must undergo a serum pregnancy test with negative result at screening and must be willing to use effective and reliable method of contraception for at least 12 months after the last satri-cel infusion. Egg donation should be refrained for 12 months.

     13. Male part

     Exclusion Criteria:

  <!-- -->

  1. The time interval between leukapheresis and completion of adjuvant chemotherapy is more than 12 weeks.
  2. Participants with high risk of bleeding, perforation or obstruction, including but not limited to deep or large ulcer, unstable/active ulcer, active or history of digestive tract bleeding/perforation/obstruction within three months.
  3. Participants who have received any non-standard adjuvant anti-tumor treatment for G/GEJ adenocarcinoma allowed in this trial, including any systemic anti-tumor drugs not specified in the protocol, any radiotherapy or interventional therapy, etc.
  4. Participants who have received systemic anti-tumor treatment for G/GEJ adenocarcinoma within 2 weeks (or within 5 half-lives of the drug, whichever is shorter) prior to leukapheresis.
  5. Participants who have received major surgery (excluding cataract surgery and others requiring local anesthesia) within 4 weeks prior to leukapheresis or significant traumatic injury and have not recovered adequately from the toxicity and/or complications. Participants who are anticipated to need major surgery during the trial will also be excluded.
  6. Participants who have received any prior genetic engineering modified cellular therapy (such as CAR T-cell, TCR T-cell, etc.).
  7. Participants with AEs from previous treatment who have not recovered to Grade ≤ 1 per Common Terminology Criteria for Adverse Events (CTCAE) v5.0, excluding hair loss, neuropathy, other events that are unlikely to cumulate toxicity from trial treatment as determined by the investigator, and laboratory abnormalities allowed in this trial.
  8. Participants with serologically positive human immunodeficiency virus (HIV), Syphilis, and hepatitis C virus (HCV). HCV antibody positive but HCV RNA negative can be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, type, and severity of adverse events | Signed ICF to 15 years after CT041 infusion
  ncidence, type, and severity of adverse events, including
  * Adverse Events (AEs)
  * Adverse Events of Special Interest (AESIs)
  * Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Disease-free survival (M12-DFS) | 12 months after surgery
  Disease-free survival (M12-DFS) rate at 12 months after surgery
Disease-free survival (DFS) after surgery | Up to approximately 24 months
  Disease-free survival (DFS) after surgery
Distant metastasis-free survival (DMFS) after surgery | Up to approximately 24 months
  Distant metastasis-free survival (DMFS) after surgery
Overall Survival (OS) | Up to approximately 24 months
  Overall Survival (OS)
To evaluate the cellular metabolism kinetics of satri-celrea under the curve (AUC) and sustained cell survival (Tlast) after satri-cel infusion | up to 18 months
  CAR copy number, time to peak amplification (Tmax), peak amplification (Cmax), area under the curve (AUC) and sustained cell survival (Tlast) after satri-cel infusion
To evaluate the immunogenicity of satri-cel | up to 18 months
  Anti-drug antibody (ADA) positive rate after infusion of satri-cel cells

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Gaobo Hospital, Beijing, Beijing Municipality
  - Nanjing Gulou Hospital, Nanjing, Jiangsu